CLINICAL TRIAL: NCT02738619
Title: Vitamin D Supplementation as an Adjuvant Therapy for Specific Immunotherapy in Patients With Allergic Rhinitis.
Brief Title: Allergic Rhinitis, Immunotherapy and Vitamin d
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, GUILLERMO VELAZQUEZ SAMANO, dr, Hospital General de Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DI/15/309/04/042
Record Dates: First submitted 2016-04-06; First posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Allergy
Keywords: allergic rhinitis; immunotherapy; vitamin D
MeSH Terms: conditions — Hypersensitivity; Rhinitis, Allergic | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin d3 (Active Comparator): 1600 UI
  Interventions: Drug: Vitamin D3
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Vitamin D3 — 1600 UI
  Other Names: vitamin d
  Arms: vitamin d3
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
Vitamin D as adjuvant to subcutaneous specific immunotherapy in patients with allergic rhinitis Specific allergen immunotherapy is the treatment of choice for patients with persistent allergic rhinitis. Some strategies to accelerate immunological and clinical changes to ensure an early response and improve adherence are needed. The administration of vitamin D along with conventional treatments in allergic patients with asthma or atopic dermatitis, pathophysiological entities like allergic rhinitis, reduces the severity of symptoms in less time.

Primary endpoint. To evaluate the efficacy of vitamin D in terms of reducing the time of therapeutic response to subcutaneous specific allergen immunotherapy.

Compare the time of clinical improvement and adherence to treatment among the group receiving vitamin D against the group receiving placebo Analyze the relationship between vitamin D values, total serum IgE, serum eosinophil and nasal cytology in both groups before and after treatment Assess the safety of vitamin D by serum calcium. TH17 and Treg quantify cells before and after treatment. MATERIAL AND METHODS This is a interventional, prospective clinical trial randomized placebo-controlled, double-blind study including paediatric patients (children 3-12 yr old) with allergic rhinitis, with parallel group: Immunotherapy + Placebo and Immunotherapy + Vitamin D. Patients prior informed consent include more patients being female and male of 3 to 12 years old. They will be randomized and in the same proportion. The sample was calculated using the G Power program to achieve an effect size of 0.65, with alpha = 0.05, statistical power = 80% and 20% losses to mean difference of 2 independent groups, the result was 80 patients, 40 per group. Monitoring will be conducted at 0, 3 and 6 months, assessing clinical and laboratory parameters with the questionnaire RQLQ, TNSS, CARACT KIDS, ARIA, GINA.

ANALYSIS It will be analyzed in SPSS. The results are expressed by descriptive statistics. For comparison of means will be used t student. It will be analyzed with ANOVA, variance for repeated measures in time, general linear model, structural equations, multivariate analysis, analysis of the main components. P values <0.05 were considered statistically significant.

DETAILED DESCRIPTION:
Vitamin D as adjuvant to subcutaneous specific immunotherapy in patients with allergic rhinitis BACKGROUND Allergic diseases are considered the pandemic of the 21 century. Allergic rhinitis (AR) is the most common with an overall prevalence of 4 to 40% in the world. In Latin America, it is a common chronic disease, with an overall prevalence in 8 countries assessed 6.6%. However, the percentage is remarkably lower than that found in ISAAC, which showed a prevalence of 27.9% in patients aged 6 to 7 years and 37.6% in 13 to 14 years. In children under 10 years, the prevalence of 11.6% in Mexico and in children aged 13 to 14 years in Mexico is 15%. Studies in Mexico, with the measuring instrument ISAAC Phase III study, reported an overall prevalence of allergic rhinitis 4.6%. Allergic rhinitis is a chronic inflammatory disease of the nasal mucosa mediated by IgE antibodies specific allergen, with the participation of various cells, cytokines, chemoattractants and mediadores. Allergic rhinitis generates direct and indirect costs including treatment of chronic disease, comorbidities, social and employment impact and escolar absenteeism. The base immunopathological allergic rhinitis is type I hypersensitivity mediated immunoglobulin type E (IgE) specific to a previously sensitized antigen, usually inhalado. Allergic sensitization and response occur in two steps. The first is the antigen uptake by antigen presenting cells (APCs) that can be professional, B lymphocytes or dendritic cell CPA. The CPA, after processing the antigen inside and present on their surface receptors with major histocompatibility complex (HLA) class II, contact a T-collaborator CD4 + (TH2) cell. This activates the TH2 cell interaction, resulting in the release of several cytokines, such as interleukins 4, 5, 9 and 13, which stimulate more TH2 cells, eosinophils and cause the differentiation of specific B cells into plasma cells producing specific immunoglobulin E against allergen. Thus large amounts of specific IgE to the blood are released. These specific IgE adhere to their receptors present high and low affinity on the surface of mast cells (also called mast cells), rendering them "sensitized". The second step is a subsequent exposure to the allergen which binds to membrane IgE producing degranulation of mast cells and release of preformed mediators such as histamine, and de novo synthesis of other mediators, including leukotrienes, prostaglandins, thromboxanes, kinins and proteasas. This response early phase of the allergic reaction occurs 10 to 30 minutes after exposure to allergens. It is useful, practical and recommended follow international guidelines ARIA (Allergic Rhinitis and Its Impact on Asthma) for the diagnosis, classification and treatment of rhinitis alérgica. ARIA proposes to investigate and analyze the clinical findings of the interrogation and physical examination such as watery rhinorrhea, congestion, obstruction and nasal itching, sneezing, allergic shiners, allergic salute, Dennie Morgan lines; and laboratory data as serum eosinophilia, serum total IgE levels increased in the absence of parasitosis and eosinophils present in the nasal cytology, it allows us to confirm the diagnosis of allergic rhinitis and its subtypes, as well as other types of rhinitis. The definitive diagnosis is made by identifying the signs, symptoms and laboratory data previously mentioned the identifiación of IgE specific to the allergen or allergens previously sensibilizado. There are two ways to identify an allergen skin tests and other blood with ImmunoCAP®. Once the definitive diagnosis of allergic rhinitis, management begins with the advice and education for the patient and his family confirmed about the disease and its treatment. Initial measures taken to prevent or mitigate the symptoms of allergic rhinitis is two; First, avoid contact with allergens triggers and second change their environment. The medium-environmental measures often include modifying factors that are known by the patient or are potentially a source of allergic response in areas such as home, school and laboral environment. Drug treatment for allergic rhinitis is with oral antihistamines and topical, oral and topical steroids, leukotriene inhibitors, membrane stabilizing mast cells, limited and controlled application of topical decongestants and anticolinérgicos. The unifying action among these drugs is modulation of the immune response to the allergen. In some cases, the pharmacological agent is specific therapeutic targets (membrane stabilizing mast cells, antihistamines) and in others, the agent has a generalized mode of action in alleviating the immune response (steroids). Skin tests allow to establish which specific allergens are causing the hiperreactividad. This is necessary before starting immunotherapy, which is administered and advised when dealing with a patient with persistent allergic rhinitis and the measures described above are insufficient to control. Documenting specific allergen sensitivity by, preferably with skin testing in vivo IgE, can route the inmunoterapia. Subcutaneous immunotherapy involves injecting staggered amounts of allergen until a "maintenance dose" or the maximum tolerated dose that relieves síntomas13. The only treatment that has succeeded in changing the natural history of disease is specific immunotherapy (SIT) with allergens; today is the treatment of elección14. Subcutaneous immunotherapy has a history of over a hundred years since its first application in England in 1911 by Leonard Noon15. It is applied in two phases: a phase of tolerance induction and maintenance. After the induction phase of tolerance in which the dose is gradually rises to reach the scheduled dose mantenimiento13 phase begins. The maintenance dose is delivered every two to six weeks, depending on the characteristics of extracto14. Immunotherapy is typically continued for three to five years and results in immunological tolerance (defined as the absence of specific immune response against an allergen, whether self or foreign, induced by previous contact) and control symptoms long term, even after suspend, up to 75% of pacientes13,14. The time it takes to start the therapeutic response is prolonged, an average of 6 meses13,14. The main drawback, as a result of this problem, poor adherence to treatment, therefore it is necessary to find strategies to accelerate the response terapéutica16. Today it is clearly known that asthma using vitamin D plus immunotherapy decrease symptoms and medication use associated with increased IgG4, IL10, TGF-b17 and T lymphocytes reg18. Also it inhibits immunological reactions such as increased cytokine profile TH17 and decreased IL-10, mediated by TH1 lymphocytes and TH 1719. In addition reduces inflammation and cytokine-mediated expression TH219 cells. Previously, in an animal model it demonstrated that vitamin D decreases IL-5 and IL-13 in 3 months20. Several estudios21,22,25, show that vitamin D stimulates the production of CD4 + CD25 + FOXP3 Treg +, which would help produce more temprano21 immunological tolerance. In patients with asthma who received immunotherapy more vitamin D compared with another group receiving only immunotherapy improvement of symptoms was documented earlier in the first group, with a statistically significativa21. Clinical trials have proven vitamin D in allergic diseases like allergic rhinitis and asthma and dermatitis atópica22. It is known that vitamin D supplementation more conventional treatment in atopic dermatitis improves the resolution of the severity of symptoms 40% faster than when conventional treatment is used alone, ie avoid the allergen, skin hydration, antihistamines and steroids; also it normalizes patterns of TH1, TH2, TH17 and Treg in 3 months22. The American Society of endocrinology considered normal serum 25 (OH) D when they are above 30 ng / ml, failure between 21 and 29 ng / ml and less than 20 ng / ml23 deficiency. Previous studies recommend that patients benefit from the additional administration of vitamin D are those exhibiting serum 25 (OH) D less than 30 ng / ml24,25. The requirements in children aged 0 to 1 year old are at least 400 IU / day and children over 1 year, at least 600 IU / day.27. To keep blood levels greater than 30 ng / ml are needed at least 1000 IU / day for children older than 1 year. To correct vitamin D deficiency values between 1000 IU and 4000 IU are used in children without graves27 problems arise. If values greater than 5000 IU in children are used estricta27 medical supervision is recommended. The side effects are alterations in serum levels of calcium and parathormona27.

PROBLEM Allergic rhinitis represents a global public health problem. In Mexico, the prevalence ranges from 10 to 30%. Immunotherapy is the treatment of choice, however, the time it takes to start the therapeutic response is prolonged, on average 6 months, which results in poor adhesion ranging from 13% to 89%. So you need to find strategies to accelerate the therapeutic response. It is known that the administration of vitamin D immunotherapy in allergic diseases, decreases symptoms as well as the use of drugs associated with increased IgG4, IL10, TGF-b and T reg cells. Also inhibits mediated immune reactions TH1 and TH17 cells the, reduces allergic inflammation and cytokine expression mediated by TH2 cells, although it is unknown whether the start time decreases action of specific immunotherapy in children with allergic rhinitis. It is known that adding vitamin D to conventional treatment of patients with atopic dermatitis decreases the severity of symptoms 40% faster (3 months) than with conventional treatment (5 months). Therefore we propose that the administration of vitamin D more immunotherapy adjuvant, may decrease the time of onset of immunotherapy at least 40% and therefore its effectiveness is improved by a better adherence.

JUSTIFICATION School and work problems experienced by patients with RA are caused by hyaline rhinorrhea, nasal obstruction and itching and sneezing in saves repetition. Often they accompanied by respiratory symptoms, such as red eye eye, eye pruritus, lacrimation and photophobia. To a lesser extent otic and palatal pruritus. Poor control of this disease is associated with poor quality of life, poor performance of daily activities in the workplace and / or study, social and economic problems. You can complicate the course of other allergic diseases .; 80% of patients with asthma suffer from allergic rhinitis and 20 to 40% of patients with allergic rhinitis are likely to have asthma. Mortality is low but morbidity is a global public health problem. Another problem of patients with rhinitis alégica is the lack of adherence to the subcutaneous specific allergen immunotherapy. It based on recent studies of well-known mechanisms of activity of vitamin D in particular elements of the immune system, and its influence on the course of allergic rhinitis this research is proposed considering the possibility of a very good simple, economic contribution and secure better adhesion of specific immunotherapy.

HYPOTHESIS If the administration of conventional treatment plus vitamin D in patients with atopic dermatitis and asthma-like allergic rhinitis entities, decreases the severity of symptoms 40% faster compared with conventional treatment, then administer vitamin D along with immunotherapy in children with allergic rhinitis will decrease at least 40% the time of onset of action of subcutaneous specific immunotherapy by earliest immunological changesTregTh17) and is consistent with standardization in laboratory values and clinical improvement assessed by questionnaires validated quality of life.

OBJECTIVES GENERAL

• Evaluate the effectiveness of vitamin D as an adjunct to specific allergen immunotherapy in children aged 5-13 years old diagnosed with allergic rhinitis in terms of reducing the time of therapeutic response.

SPECIFIC

* Compare the time of clinical improvement and adherence to treatment among the group receiving vitamin D against the group receiving placebo.
* Analyze the relationship between the values of vitamin D, serum total IgE, serum eosinophil and nasal cytology in both groups before and after treatment.
* To assess the safety of vitamin D in serum calcium in the intervention group.
* Quantify TH17 and Treg cells before and after treatment. Assess in situ expression of markers by analysis of messenger RNA transcripts Patients female and male of 5-13 years attending the General Hospital of Mexico "Dr Eduardo Liceaga" in the service of Allergy and Inmnulogía Clinic, diagnosed with allergic rhinitis, which meet the diagnostic ARIA criteria and are sensitized to a aeroallergen cutáneas28 identified by tests.

CALCULATION OF SAMPLE SIZE

In order to calculate the sample size, we rely on a study conducted in Italy and the United States on the use of vitamin D in children with atopic dermatitis. They used vitamin D plus conventional therapy. We calculated the effect size for this study was 0.65. The sample was calculated using the G Power program mean difference of 2 independent groups with als sigjuientes considerations:

Effect size = 0.65 Alpha = 0.05 Underpowered = 80% Losses = 10% The result was 80 patients, 40 per group. PROCESS

Patients 5-13 years female and male, signature of consent include prior informed consent more by their legal representatives and themselves. To meet the exclusion criteria will carry out a clinical and laboratory analysis established to assess primary and secondary immunodeficiencies, physical examination and radiography of paranasal sinuses to rule out chronic nasal pollinosis will be made, if not respond well to treatment ask tomography sinus, are excluded if they are in the service plan surgical ENT, they must be virgin of any treatment with vitamin D and have not received in the last 5 years immunotherapy for allergic diseases. They will be randomized and in the same proportion, obtained by random numbers in Excel. 3 clinical assessments and sampling for laboratory studies, baseline, another at 3 months and the last 6 months in the 2 groups will be made. clinical parameters were assessed with validated questionnaire RQLQ samples for BH, IgE, IgG, total IgA, nasal cytology were taken, skin tests with allergens based on the standards of the American Association of Alergia26 be made, serum vitamin levels are measured D. concentrations of IL-2, IL-4, IL-6, IL-10, IL-17A, IFN-γ and TNF (BD CBA Human Th1 / Th2 / Th17 Kits) shall be gauged; percentages and absolute numbers of Treg cells (CD4 + CD25 + FoxP3 +) and Th17 (CD3 + CD4 + CD161 + CD196 + (CCR6 +)). After processing the blood samples and obtain cells in the laboratory according to the suppliers recomendciones be marked with the following fluorescent antibody:

anti-CD196 (CCR6) AlexaFluor 647 anti-CD3 APC / Cy7 anti-CD4 PE-Cy5 anti-CD161 PE / Cy7 antiCD Alexa Fluor 488-25 PE anti-FoxP3 The analysis will be performed at the Research Unit Experimental Medicine, UNAM, in the laboratory HIPAM (liver, pancreas and motility). FACSCalibur flow cytometer with DIVA software II is used. at least 10,000 10,000 regulatory T cells and Th17 be analyzed.

STATISTIC ANALYSIS It will be analyzed in SPSS. The results are expressed by descriptive statistics. For comparison of means will be used t student. It will be analyzed with ANOVA, repeated measures over time and the general linear model. Additionally structural equation modeling and analysis of the main components will be made. P values <0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients female and male of 5-13 years diagnosed with persistent allergic rhinitis according to ARIA guide
2. To sign the consent and legal representatives informed consent and patient.
3. Being sensitized to a aeroallergen and are candidates for specific immunotherapy.
4. Let them bring serum levels of 25 (OH) D less than 30 ng / ml
5. are in Stage 1 or 2 Tanner.
6. BMI within the normal range (between 5 and 85 percentiles)

Exclusion Criteria:

1. primary and / or secondary immunodeficiencies
2. Chronic nasal polyposis
3. Adenoiditis and / or tonsillitis candidates for surgical resolution
4. have taken vitamin D in the last 6 months.
5. have used specific allergen immunotherapy in the last 5 years.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Rhino-conjunctivitis Questionnaire (symptom severity) | Time Frame: Baseline
  Rhino-conjunctivitis Questionnaire (symptom severity) [ Time Frame: Baseline ] [ Designated as safety issue: No ] 10cm visual analogue scale used in a 28-item questionnaire to evaluate their symptoms severity.
Rhino-conjunctivitis Questionnaire (symptom severity) | Time Frame: 3 months after intervention
  Rhino-conjunctivitis Questionnaire (symptom severity) [ Time Frame: 3 months after intervention ] [ Designated as safety issue: No ] 10cm visual analogue scale used in a 28-item questionnaire to evaluate their symptoms severity.

CONTACTS AND LOCATIONS:
Overall Officials: joselin hernandez, dr, Study Director — Hospital General de Mexico
Locations (1):
- Juan Carlos Fernandez de Cordova Aguirre, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes